CLINICAL TRIAL: NCT04235764
Title: Ex-Vivo Trial of En-bloc Transurethral Resection of Bladder Tumor (En-bloc TURBT) Specimens Using a Redesigned Surgical Resectoscope Device
Brief Title: En-bloc Transurethral Resection of Bladder Tumor (En-bloc TURBT) Specimens Using a Redesigned Surgical Resectoscope Device
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200020; 20-C-0020
Record Dates: First submitted 2020-01-18; First posted 2020-01-22 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11-13

CONDITIONS: Bladder Cancer
Keywords: TURBT; Transurethral Resection of Bladder Tumors; Cystectomy; Modified Resectoscope; Natural History
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/ Cohort 1: Bladder Cancer Patients
  Interventions: Device: modified resectoscope; Procedure: TURBT

INTERVENTIONS:
Device: modified resectoscope — The modified resectoscope will be used post cystectomy (En-bloc TURBT) to resect areas of the tumor from the cystectomy specimen. These resected tumors will be sent for histopathology to assess the size of resection, depth of resection, and ability to ascertain tumor orientation and compared to the remainder of the cystectomy specimens to see if the modified resectoscope can provide improved pathologic standards for the TURBT procedure.
Procedure: TURBT — All patients will receive routine surgical transurethral resection of bladder tumors (TURBT).

SUMMARY:
Background:

Bladder cancer is the sixth most common cancer in the United States. The way that doctors remove tumors in bladder surgeries may leave some cancer . Also, many people have their tumors return or progress after surgery. Researchers want to test a modified device. It might tell doctors more about bladder tumors.

Objective:

To see if using a modified standard device with bladder surgery can provide better information about tumors in bladder specimens.

Eligibility:

People ages 18 and older who need to have their bladder removed at the NIH.

Design:

Participants will be screened with:

Medical and prior surgical history

Review of existing MRI, x-ray, or CT scans

Review of existing specimens and reports

Pregnancy test for women of childbearing age

CT or MRI: Participants will lie in a machine. The machine will take pictures of their body.

Participants will have bladder surgery. This will occur in the same way as if they did not take part in this study. A member of the research team will cut the removed bladder using the modified device. This will most likely be done on a separate back table in the operating room. The bladder and samples after cutting will be sent out for review. The will occur just as it would if the participants were not in this study. The only difference is the way that the specimen is prepared for review.

Participants follow-up care will occur per standard of care. Or it will occur as part of any other study in which they might also be enrolled.

DETAILED DESCRIPTION:
Background:

* Bladder cancer is the sixth most common cancer in the United States, disproportionately affecting more men than women.
* The gold standard for the surgical treatment and diagnosis of non-muscle invasive bladder cancer is transurethral resection of bladder tumors (TURBT).
* TURBT requires the fragmentation of bladder tumors and piecemeal removal of these tumors.
* TURBT leads to loss of histopathologic information - including tumor orientation, size, and margin status - which may compromise outcomes and risk tumor seeding within the bladder.
* Given these multiple problems with TURBT we are testing some modifications to the current resectoscope device and the effect of these modifications on the quality of TURBT specimens produced.
* The redesigned resectoscope device will be tested ex-vivo on cystectomy specimens to avoid risks to patient safety.

Objectives:

The primary objective of this study is to determine if resectoscope device modification can provide improved pathologic standards for the TURBT procedure. An improvement in any of the parameters outlined below will constitute a device improvement in the current resectoscope:

* Presence of three tissue layers within the tumor specimens containing bladder mucosa, lamina propria, and portions of the muscularis.
* Information regarding tumor margin, assessed as the ability to ascertain if tumor is present at the margin of the resection.

Eligibility:

* Medical condition requiring surgical removal of the bladder
* Men and women, age >= 18 years

Design:

* Preclinical tissue acquisition trial, ex vivo, proof-of-concept.
* Following cystectomy, a modified resectoscope/redesigned resectoscope will be used to resect areas of tumor from the cystectomy specimens. These resected tumors will be sent with the cystectomy specimen for histopathology to assess the size of resection, depth of resection, and ability to ascertain tumor orientation.
* The remainder of the cystectomy specimens will undergo traditional histopathology. Histopathologic information from both specimens will be included in the final histopathologic diagnosis to ensure accurate oncology staging.
* This study will allow for about 2 years of accrual and the accrual ceiling will be set at 25 subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients requiring surgical removal of the bladder at the NIH Clinical Center.

NOTE: Reasons for need for surgical removal of bladder include cancer or benign condition for which a surgeon determined surgical removal of the bladder is recommended. Patient's with invasive bladder cancer requiring cystectomy are eligible for enrollment. Bladder cancer remains the most common reason for cystectomy. Patients with clinical advanced disease and having other treatments/or participating in other trials remain eligible for enrollment in this study.

* Men and women
* Age greater than or less than 18 years
* Deemed clinically appropriate for the planned surgical procedure.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Subjects will be asked to co-enroll in 15-C-0087, "Care of the Urothelial Cancer Patient and Prospective Collection of Biospecimens from Healthy Volunteers and Urothelial Cancer Patients." NOTE: Most participants are expected to already be enrolled in 15-C-0087 prior to entry in this study.

EXCLUSION CRITERIA:

- Cystectomy during pregnancy would subject the fetus to significant risk of miscarriage or premature labor. For this reason, pregnant women are ineligible for this study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bladder Cancer Patients
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of resectoscope device modification on pathologic standards for the TURBT procedure | Time of surgery/pathologic assessment (7-10 days)
  -Presence of three tissue layers with in the tumor specimens containing bladder mucosa, lamina propria, and portions of the muscularis.-Information regarding tumor margin, assessed as the ability to ascertain if tumor is present at the margin of the resection.

SECONDARY OUTCOMES:
Assessment for possible bladder perforation in bladder specimens | Time of surgery/pathologic assessment (7-10 days)
  The rate of occurrence will be described/tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Raju R Chelluri, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-C-0020.html